CLINICAL TRIAL: NCT06532370
Title: Implementing a Contingency Management Program Addressing Methamphetamine Use For and With the People of Hawaii
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's Medical Center (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RA-2024-019; U54GM138062 (NIH)
Record Dates: First submitted 2024-07-29; First posted 2024-08-01 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Contingency Managment; Methamphetamine Use Disorder

STUDY DESIGN:
Intervention Model Description: Participants will all be assigned to the CM intervention group and will be asked to follow-up three times per week for a total of 12-weeks to engage in the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Contingency Managment (Experimental): Participants are allowed to complete CM three times per week for the maximum of 12-weeks. At the six- and 12-week time points, participants will complete the Treatment Effectiveness Assessment (TEA) with study personnel.
  Interventions: Behavioral: Contingency Managment

INTERVENTIONS:
Behavioral: Contingency Managment — If the sample be methamphetamine negative, participant will be positively reinforced and offered incentives. Participants immediately draw the reinforcement slip of paper to receive a prize from a selection kept on-site. Approximately, half of the slips offer written praise (e.g. "great job!"). The other half of slips are then divided between low value (e.g. food gift cards, bus passes), medium value (e.g. prepaid cell phone, clothing gift cards), and a few large value rewards (e.g. iPad, jewelry). Should the sample be positive for methamphetamine, no reinforcement and/or incentive to be provided. Participant will be encouraged to continue to participate in CM program and follow-up on the next CM date.

SUMMARY:
The goal of this clinical trial is to use contingency management (CM) as an intervention tool to address methamphetamine use.

The main objectives are to:

* Gather effectiveness data on a pilot a CM program for participants in Hawaii who use methamphetamine following hospitalization due to traumatic injury
* To assess participant perspectives on engaging with a CM program based at a Level 1 Trauma Center. Researches will assess both patient-reported and biologically-confirmed medium-term program effectiveness and conduct qualitative interviews with participants post-program.

Participants will:

* Visit a follow-up clinic up to three times per week to complete urinalysis following discharge from the trauma unit
* Complete Treatment Effectiveness Assessments at 6 and 12-weeks
* Engage in a qualitative interview at the end of the CM program

ELIGIBILITY:
Inclusion Criteria:

* Admitted trauma patients
* Age greater than 18 years old
* Urine drug screen positive for methamphetamines during the current hospitalization
* Report at least weekly methamphetamine use
* First methamphetamine use greater than 6 months prior to injury
* Report at least 4 DSM-V Amphetamine-Type Substance Use Disorder symptoms (at least moderate disease)
* Glasgow Coma Scale ≥13 upon arrival to the emergency department
* Ability to understand and participate in study procedures
* Ability to communicate in English

Exclusion Criteria:

* Active psychosis (reporting auditory or visual hallucinations)
* Under ongoing cardiorespiratory monitoring
* Evidence of moderate or severe traumatic brain injury
* Patients who are known to be pregnant
* Prisoner
* Individuals incarcerated at the time of their hospitalization
* Individuals lacking capacity to provide, or are otherwise unable or unwilling to provide written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-10-10 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
TEA Outcomes at 6 and 12-weeks | From enrollment to 6 and 12-weeks
  Treatment Effectiveness Assessment (TEA): This assessment asks individuals to respond to changes in four domains following a drug treatment program: substance use, health, lifestyle, and community. The score for each domain can range from 1 (no change or not much) to 10 (much better), for a total score of 4-40. This score allows for the prioritization of each participants values, and therefore does not require strict abstinence to demonstrate benefit from drug treatment.

SECONDARY OUTCOMES:
Qualitative Outcomes | At the end of treatment at 12-weeks
  Interviews will be conducted as semi-structured interviews using a priori interview guides. Interviews will be transcribed and analyzed using a Template Analysis approach. Two coders will conduct coding of the interview data to ultimately identify themes that will be used as the basis for interpretation. The final analysis of the qualitative data will include contrasts and comparisons made across interviews to examine overlaps and divergences across any relevant sub-samples (e.g., sex, age). Results will present thematic patterns, how frequently each code occurs, and any contradictory evidence.

OTHER OUTCOMES:
Urine Analysis Results | From enrollment to the end of treatment at 12-weeks
  Study personnel will ask participant to complete a urine analysis screen. Following completion of the urinalysis, study personnel will use a test strip to determine if the sample is methamphetamine negative or positive. Results will be documented and analyzed for a reduction in methamphetamine.

CONTACTS AND LOCATIONS:
Overall Officials: Todd Seto, MD, Study Chair — The Queens Medical Center
Locations (1):
- The Queen's Medical Center, Honolulu, Hawaii, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gold MS, Kobeissy FH, Wang KK, Merlo LJ, Bruijnzeel AW, Krasnova IN, Cadet JL. Methamphetamine- and trauma-induced brain injuries: comparative cellular and molecular neurobiological substrates. Biol Psychiatry. 2009 Jul 15;66(2):118-27. doi: 10.1016/j.biopsych.2009.02.021. Epub 2009 Apr 5. PMID 19345341
- [Background] El Moheb M, Herrera-Escobar JP, Breen K, Orlas C, Haynes AN, Levy-Carrick NC, Nehra D, Sanchez SE, Salim A, Velmahos G, Kaafarani HMA. Long-term outcomes of psychoactive drug use in trauma patients: A multicenter patient-reported outcomes study. J Trauma Acute Care Surg. 2021 Feb 1;90(2):319-324. doi: 10.1097/TA.0000000000003032. PMID 33264267
- [Background] Ronsley C, Nolan S, Knight R, Hayashi K, Klimas J, Walley A, Wood E, Fairbairn N. Treatment of stimulant use disorder: A systematic review of reviews. PLoS One. 2020 Jun 18;15(6):e0234809. doi: 10.1371/journal.pone.0234809. eCollection 2020. PMID 32555667
- [Background] Ling W, Nadipelli VR, Solem CT, Farabee D, Ronquest NA, Perrochet B, Learned SM, Deshpande CG, Heidbreder C. Measuring recovery in opioid use disorder: clinical utility and psychometric properties of the Treatment Effectiveness Assessment. Subst Abuse Rehabil. 2019 Jun 5;10:13-21. doi: 10.2147/SAR.S198361. eCollection 2019. PMID 31239805